CLINICAL TRIAL: NCT05086991
Title: AIHEMAF - P "An Innovative Healthcare Model for AF Patients" No-profit Observational Study on the Role of the Community Pharmacist and "The Pharmacy of Services" in the Case Management of Patients Suffering From Atrial Fibrillation and Being Treated With New Generation Oral Anticoagulants
Brief Title: AIHEMAF - P "An Innovative Healthcare Model for AF Patients"
Acronym: AIHEMAF - P
Status: Completed | Type: Observational
Sponsor: Farmacia La Regina s.r.l. (Other)
Collaborators: Istituto Superiore di Sanità (Other); Università degli Studi di Brescia (Other); Nova Biomedical Italia s.r.l. (Unknown); Health Telematic Network (Industry); Centro Studi Federfarma (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2
Record Dates: First submitted 2021-09-19; First posted 2021-10-21 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Atrial Fibrillation
Keywords: adherence; therapy; follow up; community pharmacy; pharmacist; case manager; telemedicine; pharmacy of service; pharmacological therapy check; ecg; general physician; Cardiology Specialist; Doac; Noac
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group Study: Follow up of the patients for 12 months by the community pharmacist in the role of case manager and execution of the activities foreseen by the PAI (individual assistance plan) through telemedicine (ecg, cardiac holter) and self analysis (hemoglobin, hematocrit, creatinine).
  Interventions: Other: Follow up

INTERVENTIONS:
Other: Follow up — like group descriptions

SUMMARY:
Non-profit observational study on the role of the community pharmacist and "the pharmacy of services" in the case management of patients suffering from atrial fibrillation and being treated with new generation oral anticoagulants

DETAILED DESCRIPTION:
Atrial fibrillation is one of the most common cardiac arrhythmias, from which, in Italy, more than a million people are affected and estimates speak of an increase of up to 70% in the coming years. Due to its ability to increase the thrombo-embolic risk, the affected people are subjected to anticoagulant and antiarrhythmic pharmacological interventions in order to protect the patient from highly disabling events such as cerebral stroke or other arterial embolisms.

However, these pharmacological therapies require a dynamic approach over time, as the choice of active ingredients and the relative dosages depend on the patient's overall health status and for this reason it is important that he adheres to the monitoring plan, prepared by a specialist in cardiology, so that therapeutic appropriateness is always guaranteed.ù

In daily clinical practice, the follow-up activities, defined by the guidelines of the European Society of Cardiology (ESC), consist in the evaluation of:

* General health status
* Bleeding events and related risk
* Therapeutic adherence
* Kidney function
* Drug interactions
* Control of heart rhythm and related symptoms
* Pathology progression

In the recent past, these activities were carried out solely and exclusively by the Specialist Doctor, as the only person authorized to prescribe the new oral anticoagulant drugs. Only recently, with the introduction of the AIFA 97 note, the General Practitioner was given the opportunity to prescribe these drugs to the patient suffering from Non-Valvular Atrial Fibrillation and to carry out the necessary monitoring. Consequently, the visit to the Specialist is reduced to once a year or whenever the General Practitioner deems it appropriate.

However, the recent epidemiological emergency has highlighted the need to redesign the follow-up pathways of these patients in order to reduce interpersonal contacts today and to simplify those pathways tomorrow. In fact, nowadays, patients suffering from atrial fibrillation and on anticoagulant therapy must carry out a series of interminable steps to comply with all the activities provided for in their follow-up plan. This, as the National Health System is organized today, therefore, translates into a lose-lose scenario, due to the lack of reconciliation between the diagnostic and therapeutic activities to be carried out and the rhythms of life.

On the basis of this, it is necessary to design follow-up models, which, thanks to the territorial integration of all the care settings and the related health professionals available, allow the patient to be able to enjoy 0 km assistance models, which allow him to carry out the activities provided for in the treatment plans in the simplest and most immediate way possible in order to be able to guarantee in a timely manner the most suitable treatments for your state of health, foreseeing and preventing complications and responding effectively and efficiently to the needs emerging.

Among the health professionals available to date, that of the Territorial Pharmacist is little considered, which represents, due to the position in which it is found within the National Health Service, a potential that has not yet been fully exploited. In fact, he could take on the role of case manager (professional who manages one or more cases entrusted to him according to a predetermined path, such as the PDTA, in a defined space-time context) of the patient suffering from atrial fibrillation and in therapy with oral anticoagulants of new generation thanks to the capillarity on the territory, the hourly availability higher than any other territorial health facility, the health skills in its possession and what it can offer in terms of services within the so-called "service pharmacy". In this scenario, the pharmacist would not replace any of the other actors already present in the multidisciplinary care team but would integrate into it and, moreover, being already affiliated with the National Health Service, the conferral of this role would not cause a excessive cost increases, such as that which would result from hiring new staff to achieve the same goals. The involvement of local pharmacists in the case management of these patients could represent the "sustainable" key for de-hospitalization of chronic patients, which has been talked about for some time without being able to find concrete and at the same time not particularly costly solutions, and the gateway to the Service National Healthcare that allows them to monitor their state of health, be supported in their activities and remain connected with all the other actors in the care process.

ELIGIBILITY:
Inclusion Criteria:

* age> 18 years,
* patients suffering from Non-Valvular Atrial Fibrillation and being treated with new generation oral anticoagulants;
* able to express consent to the study;
* regularly related to the trial site (Farmacia La Regina S.r.l.)
* AntiCovid19 vaccination performed.

Exclusion Criteria:

* Nobody

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients suffering from Non-Valvular Atrial Fibrillation and being treated with new generation oral anticoagulants;
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Model implementation description | 12 months
  The primary outcome is mainly descriptive. In fact, the primary objective of the study is to describe the implementation and outcomes of an innovative Smart Clinic model useful for the clinical and pharmacological monitoring of the patient suffering from non-valvular atrial fibrillation treated with new generation oral anticoagulants, in which a community pharmacist, adequately trained, takes on the role of case manager and the patient has the possibility to perform the checks provided in telemedicine and in self-analysis, in the service pharmacy regime, the results of which will be shared in real time with the treating physician and reference specialist of the same. This model is new as there is no coagulation clinic in Italy as in other countries of the world.

SECONDARY OUTCOMES:
Percent of Participants With Adherence to the PDTA | 12 months
  Measure of the variation of the percentage of adherence to PDTA (patients who performed the scheduled checks at 1-3-6-12 months / total of patients enrolled x 100) in the cohort of the patients enrolled in the study and therefore followed from a case manager identified in the community pharmacist with the opportunity to perform the checks provided in telemedicine and in self-analysis, thanks to the exploitation of "pharmacy of service".
Prescriptive appropriateness | 12 months
  detection of the number of cases in which the therapy must be changed (molecule or dosage) or suspended because it is not appropriate
Adherence to therapy | 12 months
  detection of cases in which the therapy was not followed correctly
Pharmacological problems | 12 months
  detection of cases in which drug therapy needs to be revised due to drug-drug interactions
Bleeding and / or thrombo-embolic complications; | 12 months
  detection of cases of bleeding and / or thrombo-embolic complications
Acceptance of reports | 12 months
  detection of cases in which the general practitioner or specialist doctor accepts the reports of the pharmacist
Economic Impact | 12 months
  Evaluation of the economic impact secondary to the establishment of the figure of the community pharmacist as Case Manager and to the use of the "pharmacy of service" (Comparison costs/benefits in euro between traditional assistence model and this innovative assistance model) (comparison between the costs currently incurred by the Italian health care system for the assistance to AF patients on doac therapy and the related benefits and costs deriving from the adoption of a care model such as the one object of research and the relative benefits)

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele La Regina, DR, Principal Investigator — Farmacia La Regina srl
Locations (1):
- Farmacia La Regina s.r.l., San Rufo, Salerno, Italy

IPD SHARING:
Plan to Share IPD: No
The data will be shared only in aggregate and anonymous form.

REFERENCES:
- [Background] Corrigendum to: 2020 ESC Guidelines for the diagnosis and management of atrial fibrillation developed in collaboration with the European Association of Cardio-Thoracic Surgery (EACTS). Eur Heart J. 2021 Feb 1;42(5):546-547. doi: 10.1093/eurheartj/ehaa945. No abstract available. PMID 33242070
- [Background] Steffel J, Verhamme P, Potpara TS, Albaladejo P, Antz M, Desteghe L, Haeusler KG, Oldgren J, Reinecke H, Roldan-Schilling V, Rowell N, Sinnaeve P, Collins R, Camm AJ, Heidbuchel H; ESC Scientific Document Group. The 2018 European Heart Rhythm Association Practical Guide on the use of non-vitamin K antagonist oral anticoagulants in patients with atrial fibrillation. Eur Heart J. 2018 Apr 21;39(16):1330-1393. doi: 10.1093/eurheartj/ehy136. PMID 29562325
- [Background] Barnes GD, Sippola E, Dorsch M, Errickson J, Lanham M, Allen A, Spoutz P, Sales AE, Sussman J. Applying population health approaches to improve safe anticoagulant use in the outpatient setting: the DOAC Dashboard multi-cohort implementation evaluation study protocol. Implement Sci. 2020 Sep 21;15(1):83. doi: 10.1186/s13012-020-01044-5. PMID 32958020
- [Background] Sylvester KW, Ting C, Lewin A, Collins P, Fanikos J, Goldhaber SZ, Connors JM. Expanding anticoagulation management services to include direct oral anticoagulants. J Thromb Thrombolysis. 2018 Feb;45(2):274-280. doi: 10.1007/s11239-017-1602-1. PMID 29274044
- [Background] Andreu Cayuelas JM, Caro Martinez C, Flores Blanco PJ, Elvira Ruiz G, Albendin Iglesias H, Cerezo Manchado JJ, Bailen Lorenzo JL, Januzzi JL, Garcia Alberola A, Manzano-Fernandez S. Kidney function monitoring and nonvitamin K oral anticoagulant dosage in atrial fibrillation. Eur J Clin Invest. 2018 Jun;48(6):e12907. doi: 10.1111/eci.12907. Epub 2018 Apr 22. PMID 29423910
- [Background] Fava JP, Starr KM, Ratz D, Clemente JL. Dosing challenges with direct oral anticoagulants in the elderly: a retrospective analysis. Ther Adv Drug Saf. 2018 May 17;9(8):405-414. doi: 10.1177/2042098618774498. eCollection 2018 Aug. PMID 30364869
- [Background] Ashjian E, Kurtz B, Renner E, Yeshe R, Barnes GD. Evaluation of a pharmacist-led outpatient direct oral anticoagulant service. Am J Health Syst Pharm. 2017 Apr 1;74(7):483-489. doi: 10.2146/ajhp151026. PMID 28336758
- [Background] Kim JJ, Hill HL, Groce JB 3rd, Granfortuna JM, Makhlouf TK. Pharmacy Student Monitoring of Direct Oral Anticoagulants. J Pharm Pract. 2018 Oct;31(5):462-468. doi: 10.1177/0897190017752713. Epub 2018 Jan 24. PMID 29366379
- [Background] Li X, Zuo C, Lu W, Zou Y, Xu Q, Li X, Lv Q. Evaluation of Remote Pharmacist-Led Outpatient Service for Geriatric Patients on Rivaroxaban for Nonvalvular Atrial Fibrillation During the COVID-19 Pandemic. Front Pharmacol. 2020 Aug 21;11:1275. doi: 10.3389/fphar.2020.01275. eCollection 2020. PMID 32973511
- [Background] Miele C, Taylor M, Shah A. Assessment of Direct Oral Anticoagulant Prescribing and Monitoring Pre- and Post-Implementation of a Pharmacy Protocol at a Community Teaching Hospital. Hosp Pharm. 2017 Mar;52(3):207-213. doi: 10.1310/hpj5203-207. PMID 28439135
- [Background] Ertl J, Chalmers L, Bereznicki L. The Quality of Advice Provided by Pharmacists to Patients Taking Direct Oral Anticoagulants: A Mystery Shopper Study. Pharmacy (Basel). 2020 Sep 3;8(3):164. doi: 10.3390/pharmacy8030164. PMID 32899401
- [Background] Shimizu T, Momose Y, Ogawa R, Takahashi M, Echizen H. Impact of Pharmacists' audit on improving the quality of prescription of dabigatran etexilate methanesulfonate: a retrospective study. J Pharm Health Care Sci. 2017 Jan 17;3:4. doi: 10.1186/s40780-017-0077-8. eCollection 2017. PMID 28116115
- [Background] Virdee MS, Stewart D. Optimizing the use of oral anticoagulant therapy for atrial fibrilation in primary care: a pharmacist-led intervention. Int J Clin Pharm. 2017 Feb;39(1):173-180. doi: 10.1007/s11096-016-0419-x. Epub 2017 Jan 3. PMID 28050712

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-10-05): https://cdn.clinicaltrials.gov/large-docs/91/NCT05086991/Prot_SAP_000.pdf
  • Informed Consent Form (2021-06-16): https://cdn.clinicaltrials.gov/large-docs/91/NCT05086991/ICF_001.pdf